CLINICAL TRIAL: NCT01776528
Title: A Phase 1 Randomized, Double Blind, Placebo Controlled, Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of NGM282 in Healthy Adult Participants
Brief Title: Phase 1 SAD and MAD Study of NGM282 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 12-0101
Record Dates: First submitted 2013-01-18; First posted 2013-01-28 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — aldafermin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Cohort 1 SAD (Experimental): NGM282 Dose 1 vs Placebo
  Interventions: Biological: NGM282; Biological: Placebo
- Cohort 2 SAD (Experimental): NGM282 Dose 2 vs Placebo
  Interventions: Biological: NGM282; Biological: Placebo
- Cohort 3 SAD (Experimental): NGM282 Dose 3 vs Placebo
  Interventions: Biological: NGM282; Biological: Placebo
- Cohort 4 SAD (Experimental): NGM282 Dose 4 vs Placebo
  Interventions: Biological: NGM282; Biological: Placebo
- Cohort 5 SAD (Experimental): NGM282 Dose 5 vs Placebo
  Interventions: Biological: NGM282; Biological: Placebo
- Cohort 6 SAD (Experimental): NGM282 Dose 6 vs Placebo
  Interventions: Biological: NGM282; Biological: Placebo
- Cohort 7 MAD (Experimental): NGM282 Dose 1 vs Placebo
  Interventions: Biological: NGM282; Biological: Placebo
- Cohort 8 MAD (Experimental): NGM282 Dose 2 vs Placebo
  Interventions: Biological: NGM282; Biological: Placebo
- Cohort 9 MAD (Experimental): NGM282 Dose 3 vs Placebo
  Interventions: Biological: NGM282; Biological: Placebo
- Cohort 10 MAD (Experimental): NGM282 Dose 4 vs Placebo
  Interventions: Biological: NGM282; Biological: Placebo
- Cohort 11 MAD (Experimental): NGM282 Dose 5 vs Placebo
  Interventions: Biological: NGM282; Biological: Placebo
- Cohort 12 MAD (Experimental): NGM282 Dose 6 vs Placebo
  Interventions: Biological: NGM282; Biological: Placebo

INTERVENTIONS:
Biological: NGM282
Biological: Placebo

SUMMARY:
The purpose of this study is to determine the safety and tolerability of NGM282, both single dose and multiple doses, in normal healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, between 18 and 65 years of age, inclusive
* BMI range is 20-35 kg/m2, inclusive for the SAD Module, and 25-35 kg/m2, inclusive for the MAD Module at Screening;
* In good health, determined by no clinically significant findings from medical history, physical exam, 12 lead ECG, clinical laboratory findings, and vital signs at Screening and Day -1

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, GI, neurological, or psychiatric disorder (as determined by the PI)
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 7 days and 14 days
  To evaluate the safety and tolerability of single ascending doses and multiple ascending doses of NGM282 in healthy adult participants.

SECONDARY OUTCOMES:
Pharmacokinetics | 7 days and 14 days
  To evaluate the pharmacokinetics of single ascending doses and multiple ascending doses of NGM282 in healthy adult participants.
Pharmacodynamics | 7 days and 14 days
  To evaluate the pharmacodynamics of single ascending doses and multiple ascending doses of NGM282 in healthy adult participants.

CONTACTS AND LOCATIONS:
Overall Officials: Alex M DePaoli, MD, Study Director — NGM Biopharmaceuticals, Inc
Locations (1):
- NGM Clinical Study Site, Perth, Western Australia, Australia

REFERENCES:
- See also: Related Info — http://ngmbio.com/